CLINICAL TRIAL: NCT00567749
Title: Clinical Sensitivity of the Clearview® COMPLETE HIV 1/2, PMA # BP050009 and the Clearview® HIV 1/2 STAT-PAK®, PMA #BP050010 in the 12 - 17 Year Old Pediatric Population
Brief Title: Clinical Sensitivity of Clearview Rapid Tests in 12-17 y/o Pediatric Population
Status: Completed | Type: Observational
Sponsor: Chembio Diagnostic Systems, Inc. (Industry)
Collaborators: Inverness Medical Innovations (Industry); University of Maryland (Other); Focus Diagnostics, Inc. (Industry)
Responsible Party: Thomas D. Ippolito / VP Regulatory Affairs, Chembio Diagnostic Systems, Inc.
Other Study IDs: 02-HIV02.01
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV-1 Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A, Observational

SUMMARY:
This study is to establish the clinical sensitivity of the Chembio Diagnostics Systems, Inc. Clearview COMPLETE HIV 1/2 Assay and Clearview HIV 1/2 Stat-Pak Assay (Clearview HIV tests) in pediatric subjects who are between 12 and 17 years of age. A minimum of ten (10) known HIV-positive participants will be tested.

DETAILED DESCRIPTION:
In order to achieve the primary objective, clinical trials will be conducted to establish and confirm the sensitivity of the Clearview HIV 1/2 tests in the described pediatric population. Only HIV-1 will be included in the study.

The Clearview HIV tests can be used as a safe and effective screening method to aid in the diagnosis of infection with HIV 1/2 in the pediatric population aged between 12 and 17 years.

The secondary objectives of this study include demonstrating that:

- The Clearview HIV tests detect HIV-1 antibodies in a variety of sample matrices: capillary (fingertip) whole blood, venous whole blood, plasma and serum.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 12 years of age and no older than 17 years of age.
* Must be willing to sign (and be given) a copy of the written Information and Assent Form.
* Must have a parent or guardian present to sign and receive a copy of the Informed Consent Form.
* Must be able to provide one or two fingerstick blood samples.
* Must be able to provide three tubes of blood by venipuncture from the arm or hand only.

Exclusion Criteria:

* Have a life threatening illness (with the exception of HIV or AIDS).
* Have a suppressed immune systems (i.e. transplant patients, individuals diagnosed with non-HIV immunosuppressive illness, etc.), as determined by interviewing the study participant or parent/legal guardian.
* Have participated or are participating in a clinical trial for an HIV vaccine (as determined by interviewing the study participant or parent/legal guardian).
* Have previously participated in this clinical trial (no duplicate enrollments).
* Are currently on HAART, except as agreed on a case-by-case basis.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patient population intended for this study (study participants) consists of a minimum of 10 individuals, known to have previously tested positive for HIV antibodies, who are between 12 and 17 years of age. The patients should not be on HAART, however, the sponsor reserves the option to include a limited number of HAART patients for investigational purposes. The number of HAART patients enrolled will depend on the available pediatric HIV positive participant pool. HAART patients will be clearly identified and will be additional to the enrollment needed to meet the study objectives.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The Clearview HIV tests provide a 100% agreement with known HIV(+) status for all 10 eligible 12 to 17 year old individuals, at least one of whom will be age 12. | 3-10 days

SECONDARY OUTCOMES:
The Clearview tests will be used in a representative clinical setting for the qualitative detection of antibodies to HIV-1 in fingerstick, venous whole blood, serum and plasma matrices. | 3-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Neil T. Constantine, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Laboratory of Viral Diagnostics, University of Maryland School of Medicine, Baltimore, Maryland, United States